CLINICAL TRIAL: NCT03893227
Title: Prevalence of Nasal Hyperreactivity in Chronic Upper Airway Inflammation: a Prevalence Study
Brief Title: Prevalence of Nasal Hyperreactivity in Chronic Upper Airway Inflammation
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Laura Van Gerven, Professor doctor, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S62213
Record Dates: First submitted 2019-03-20; First posted 2019-03-28 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Hyperactivity; Chronic Rhinosinusitis (Diagnosis); Chronic Rhinitis; Upper Respiratory Disease
MeSH Terms: conditions — Spasm; Disease; Respiration Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with chronic upper airway inflammation
  Interventions: Other: Questionnaire
- Healthy control: Healthy controls without chronic upper airway inflammation
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients and healthy controls will fill out a questionnaire

SUMMARY:
Rhinitis, or inflammation of the nasal mucosa, can present with nasal obstruction, nasal discharge, itch or sneezing. If the sinusal mucosa is involved as well, it is called rhinosinusitis and facial pain or loss of smell is possible. Several causes are known, such as an underlying allergy ("allergic rhinitis", AR). If at least 2 symptoms are present for at least 12 weeks, it is called "chronic rhinosinusitis" (CRS).

Up to 2/3 of the AR and CRS patients have symptoms upon exposure to triggers such as sudden temperature changes, smoke, fragrances… a phenomenon called "nasal hyperreactivity" (NHR). It is currently not clear why some patients suffer NHR while others do not.

In this study, the investigators want to determine the prevalence and severity of nasal hyperreactivity in patients with chronic upper airway inflammation. To this end, patients and healthy controls will be asked to fill out a questionnaire inquiring presence and severity of nasal symptoms upon exposure to particular environmental triggers.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* age 18-65 y
* Nasal inflammatory symptoms for 12 weeks or longer (nasal obstruction, post-nasal drip, rhinorrhea, loss of smell, sneezing/itch, facial pain)
* Signed informed consent

Exclusion Criteria:

- Current or medical history of malignancy in the last ten years

CONTROLS

Inclusion Criteria:

* age 18-65 y
* No nasal inflammatory symptoms for 12 weeks or longer (nasal obstruction, post-nasal drip, rhinorrhea, loss of smell, sneezing/itch, facial pain)
* Signed informed consent

Exclusion Criteria:

- Current or medical history of malignancy in the last ten years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic inflammation of the upper airways. Controls without chronic inflammation of the upper airways.
Sampling Method: Probability Sample
Enrollment: 756 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the proportion of patients and healthy volunteers with nasal hyperreactivity | 3 months
  Every participant will fill out a questionnaire inquiring presence of nasal symptoms evoked by environmental triggers and lasting longer than ten minutes (nasal hyperreactivity). The proportion of patients and healthy volunteers with nasal hyperreactivity will be compared.

SECONDARY OUTCOMES:
Comparison of nasal symptom severity in patients and healthy volunteers with and without nasal hyperreactivity. | 3 months
  Every participant will fill out a questionnaire inquiring nasal symptom severity by means of a visual analogue scale (VAS). The severity of symptoms will be scored on a horizontal line of 10 cm, where 0 cm equals "no symptoms" and 10 cm equals "very severe symptoms". The VAS-scores of patients and healthy volunteers with and without nasal hyperreactivity will be compared.
Comparison of the proportion of healthy volunteers and four groups of patients (allergic rhinitis, non-allergic non-infectious rhinitis, chronic rhinosinusitis with nasal polyps, chronic rhinosinusitis without nasal polyps) with nasal hyperreactivity. | 3 months
  Every participant will fill out a questionnaire inquiring presence of nasal symptoms evoked by environmental triggers and lasting longer than ten minutes (nasal hyperreactivity). The proportion of healthy volunteers and four groups of patients (allergic rhinitis, non-allergic non-infectious rhinitis, chronic rhinosinusitis with nasal polyps, chronic rhinosinusitis without nasal polyps) with nasal hyperreactivity will be compared.
Comparison of nasal symptom severity in healthy volunteers and four groups of patients [allergic rhinitis, non-allergic non-infectious rhinitis, chronic rhinosinusitis (CRS) with and CRS without nasal polyps] with and without nasal hyperreactivity. | 3 months
  Every participant will fill out a questionnaire inquiring nasal symptom severity by means of a visual analogue scale (VAS). The severity of symptoms will be scored on a horizontal line of 10 cm, where 0 cm equals "no symptoms" and 10 cm equals "very severe symptoms". The VAS-scores of healthy volunteers and four groups of patients (allergic rhinitis, non-allergic non-infectious rhinitis, chronic rhinosinusitis with nasal polyps, chronic rhinosinusitis without nasal polyps) with and without nasal hyperreactivity will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Van Gerven, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZLeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No